CLINICAL TRIAL: NCT04037436
Title: A Model for Delivering Strength Training and Nutrition Education for Older Adults (MoveStrong): A Pilot Randomized Controlled Trial
Brief Title: Functional Exercise and Nutrition Education Program for Older Adults
Acronym: MoveStrong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); City of Lakes family Health Team (Unknown); Schlegel-UW Research Institute for Aging (Unknown); YMCA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20190401
Record Dates: First submitted 2019-06-28; First posted 2019-07-30 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2022-11

CONDITIONS: Chronic Disease; Frail; Diabetes Mellitus; Cancer; Chronic Lung Disease; Cardiovascular Diseases; Congestive Heart Failure; Hypertension; Osteoporosis, Osteopenia; Arthritis; Stroke; Kidney Diseases
Keywords: Strength Training; Balance Training; Nutrition Education; Older adults; Frailty; Feasibility
MeSH Terms: conditions — Chronic Disease; Diabetes Mellitus; Neoplasms; Cardiovascular Diseases; Heart Failure; Hypertension; Osteoporosis; Bone Diseases, Metabolic; Arthritis; Stroke; Kidney Diseases; Frailty | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: We will use a closed cohort stepped wedge design at 4 sites (1 in Northern Ontario and 3 in Southern Ontario). In a stepped wedge, sites are cluster-randomized to implement MoveSTroNg at one of four start times, each three weeks apart.
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): At regular intervals (the "steps") one cluster (i.e., one site) is randomised to cross from the control to the intervention under evaluation. This process continues until all clusters have crossed over to be exposed to the intervention. At the end of the study there will be a period when all clusters are exposed. Four sites are cluster-randomized to implement MoveSTroNg at one of four start times, each three weeks apart.
  Interventions: Other: Strength and Balance Training & Nutrition Education
- Control (Other): Each cluster contributes observations under both control and intervention observation periods.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Strength and Balance Training & Nutrition Education — Exercise:A kinesiologist-led twice-weekly program. Prior to attending the program, each attendee gets a 1:1 session with the kinesiologist to decide exercise starting levels. Group exercises start with a warm-up stepping game. Participants then perform 2 sets of 8 repetitions of each exercise, gradually progressing to an intensity of 3-8 repetitions maximum. Exercises include one each of a push, pull, squat, reach/press, lunge/step-up, lift and carry movement. After, there is a 10-minute group discussion to prompt making exercise routine at home. Nutrition:Two dietitian-led interactive group seminars to promote strategies to increase protein intake and sampling of protein-rich snacks and protein supplements. Seminar topics consider the cost to prepare high protein foods, the ability of retirement home residents to alter diet, how and why to spread protein intake through the day, how much protein is in their usual choices, and easy-to-consume protein-rich snacks.
  Arms: Intervention
Other: Usual Care — During periods when a site is not involved in the MoveSTroNg program, participants will continue with their usual care routine. Usual care routines should not involve strength and balance exercises.
  Arms: Control

SUMMARY:
There is strong evidence that specific types of exercise can improve health and physical function in older adults. While community exercise classes exist, many older adults with chronic conditions may need guidance from credentialed exercise professionals to ensure sufficient dose and progression and to address fears or low exercise self-efficacy. Furthermore, low protein intake among older adults is common and initiating exercise when nutrition is inadequate may cause weight loss and limit gains in muscle strength. The primary goal is to determine the feasibility of implementing the MoveSTroNg program under real-world conditions, measured through referral and recruitment to the program and study retention and adherence rates.

DETAILED DESCRIPTION:
The MoveStrong trial is a 1-year pilot closed cohort stepped wedge randomized control trial (RCT) to evaluate the feasibility of implementation of the MoveStrong program. This program includes a functional exercise and nutrition program that teaches older adults with chronic diseases how to perform functional resistance and balance exercises and promote adequate protein intake and nutrition. Four sites (1 Northern and 3 Southern Ontario sites) will be cluster-randomized to implement MoveStrong at one of four start times, each three weeks apart. The primary outcome will be to determine the feasibility of recruitment and referral from diverse settings (i.e., retirement homes, community centers, and family health teams) and establish the retention and adherence to the program. Secondary objectives will determine the following: What are the participant's and provider's experience with the MoveStrong program? What is the short-term responsiveness (i.e., ability to detect change) of frailty indicators (Fried Frailty Index components), protein intake, or quality of life? Who agrees to participate? What adaptations need to be made to MoveStrong, or study methods in each setting? What is the cost relative to the benefit? Is behaviour change maintained in the maintenance period? Our long term goal is to use the information from this project to develop, implement, and evaluate a sustainable, scalable and pragmatic model to deliver strength and balance training and promote adequate protein intake among older adults with chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Speak English or attend with a translator;
* ≥ 60 years;
* FRAIL scale score ≥1;
* Have ≥1 diagnosed chronic condition (i.e., diabetes, obesity, cancer (other than minor skin cancer), chronic lung disease, cardiovascular disease, congestive heart failure, hypertension, osteoporosis, arthritis, stroke, or kidney disease).

Exclusion Criteria:

* Currently doing similar resistance exercise ≥2x/week;
* In palliative care;
* Not able to perform basic activities of daily living;
* Cognitive impairment (e.g., unable to follow two-step commands);
* Travelling >1 week during exposure;
* Absolute exercise contraindications (i.e., if they select "no" to any question in the Get Active Questionnaire they must seek physician approval before exercising)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Chaplin Family YMCA, Cambridge, Ontario
  - Your Family Health Team, Greater Sudbury, Ontario
  - The Village of Arbour Trails, Guelph, Ontario
  - Village of Winston Park, Kitchener, Ontario
  - A.R. Kaufman Family YMCA, Kitchener, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
If requested we will consider sharing data. If raw data is shared, participant data will be deidentified.

REFERENCES:
- [Background] Beaudart C, Rizzoli R, Bruyere O, Reginster JY, Biver E. Sarcopenia: burden and challenges for public health. Arch Public Health. 2014 Dec 18;72(1):45. doi: 10.1186/2049-3258-72-45. eCollection 2014. PMID 25810912
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Sherrington C, Michaleff ZA, Fairhall N, Paul SS, Tiedemann A, Whitney J, Cumming RG, Herbert RD, Close JCT, Lord SR. Exercise to prevent falls in older adults: an updated systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(24):1750-1758. doi: 10.1136/bjsports-2016-096547. Epub 2016 Oct 4. PMID 27707740
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Background] Brosseau L, Wells GA, Poitras S, Tugwell P, Casimiro L, Novikov M, Loew L, Sredic D, Clement S, Gravelle A, Kresic D, Hua K, Lakic A, Menard G, Sabourin S, Bolduc MA, Ratte I, McEwan J, Furlan AD, Gross A, Dagenais S, Dryden T, Muckenheim R, Cote R, Pare V, Rouhani A, Leonard G, Finestone HM, Laferriere L, Haines-Wangda A, Russell-Doreleyers M, De Angelis G, Cohoon C. Ottawa Panel evidence-based clinical practice guidelines on therapeutic massage for low back pain. J Bodyw Mov Ther. 2012 Oct;16(4):424-55. doi: 10.1016/j.jbmt.2012.04.002. Epub 2012 Jun 23. PMID 23036876
- [Background] Giangregorio LM, Papaioannou A, Macintyre NJ, Ashe MC, Heinonen A, Shipp K, Wark J, McGill S, Keller H, Jain R, Laprade J, Cheung AM. Too Fit To Fracture: exercise recommendations for individuals with osteoporosis or osteoporotic vertebral fracture. Osteoporos Int. 2014 Mar;25(3):821-35. doi: 10.1007/s00198-013-2523-2. Epub 2013 Nov 27. PMID 24281053
- [Background] Ravindran AV, Balneaves LG, Faulkner G, Ortiz A, McIntosh D, Morehouse RL, Ravindran L, Yatham LN, Kennedy SH, Lam RW, MacQueen GM, Milev RV, Parikh SV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 5. Complementary and Alternative Medicine Treatments. Can J Psychiatry. 2016 Sep;61(9):576-87. doi: 10.1177/0706743716660290. Epub 2016 Aug 2. PMID 27486153
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Peterson MD, Sen A, Gordon PM. Influence of resistance exercise on lean body mass in aging adults: a meta-analysis. Med Sci Sports Exerc. 2011 Feb;43(2):249-58. doi: 10.1249/MSS.0b013e3181eb6265. PMID 20543750
- [Background] Borde R, Hortobagyi T, Granacher U. Dose-Response Relationships of Resistance Training in Healthy Old Adults: A Systematic Review and Meta-Analysis. Sports Med. 2015 Dec;45(12):1693-720. doi: 10.1007/s40279-015-0385-9. PMID 26420238
- [Background] Liu CJ, Latham NK. Progressive resistance strength training for improving physical function in older adults. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD002759. doi: 10.1002/14651858.CD002759.pub2. PMID 19588334
- [Background] Trombetti A, Hars M, Hsu FC, Reid KF, Church TS, Gill TM, King AC, Liu CK, Manini TM, McDermott MM, Newman AB, Rejeski WJ, Guralnik JM, Pahor M, Fielding RA; LIFE Study Investigators. Effect of Physical Activity on Frailty: Secondary Analysis of a Randomized Controlled Trial. Ann Intern Med. 2018 Mar 6;168(5):309-316. doi: 10.7326/M16-2011. Epub 2018 Jan 9. PMID 29310138
- [Background] Wang E, Keller H, Mourtzakis M, Rodrigues IB, Steinke A, Ashe MC, Thabane L, Brien S, Funnell L, Cheung AM, Milligan J, Papaioannou A, Weston ZJ, Straus S, Giangregorio L. MoveStrong at home: a feasibility study of a model for remote delivery of functional strength and balance training combined with nutrition education for older pre-frail and frail adults. Appl Physiol Nutr Metab. 2022 Dec 1;47(12):1172-1186. doi: 10.1139/apnm-2022-0195. Epub 2022 Sep 15. PMID 36108334
- [Result] Rodrigues IB, Wagler JB, Keller H, Thabane L, Weston ZJ, Straus SE, Papaioannou A, Mourtzakis M, Milligan J, Isaranuwatchai W, Loong D, Jain R, Funnell L, Cheung AM, Brien S, Ashe MC, Giangregorio LM. Encouraging older adults with pre-frailty and frailty to "MoveStrong": an analysis of secondary outcomes for a pilot randomized controlled trial. Health Promot Chronic Dis Prev Can. 2022 Jun;42(6):238-251. doi: 10.24095/hpcdp.42.6.02. PMID 35766913
- [Result] Rodrigues IB, Wang E, Keller H, Thabane L, Ashe MC, Brien S, Cheung AM, Funnell L, Jain R, Loong D, Isaranuwatchai W, Milligan J, Mourtzakis M, Papaioannou A, Straus S, Weston ZJ, Giangregorio LM. The MoveStrong program for promoting balance and functional strength training and adequate protein intake in pre-frail older adults: A pilot randomized controlled trial. PLoS One. 2021 Sep 24;16(9):e0257742. doi: 10.1371/journal.pone.0257742. eCollection 2021. PMID 34559837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Within one-week of randomization but prior to the start of the intervention, five individuals dropped out.
Groups:
- Arbour Trails; Kinnect to Wellness; Winston Park; YMCAs: At regular intervals (the "steps") one cluster (i.e., one site) is randomised to cross from the control to the intervention under evaluation. This process continues until all clusters have crossed over to be exposed to the intervention. At the end of the study there will be a period when all clusters are exposed. Four sites are cluster-randomized to implement MoveSTroNg at one of four start times, each three weeks apart.
  Strength and Balance Training & Nutrition Education: Exercise:A kinesiologist-led twice-weekly program. Prior to attending the program, each attendee gets a 1:1 session with the kinesiologist to decide exercise starting levels. Group exercises start with a warm-up stepping game. Participants then perform 2 sets of 8 repetitions of each exercise, gradually progressing to an intensity of 3-8 repetitions maximum. Exercises include one each of a push, pull, squat, reach/press, lunge/step-up, lift and carry movement. After, there is a 10-minute group discussion to prompt making exercise routine at home. Nutrition:Two dietitian-led interactive group seminars to promote strategies to increase protein intake and sampling of protein-rich snacks and protein supplements. Seminar topics consider the cost to prepare high protein foods, the ability of retirement home residents to alter diet, how and why to spread protein intake through the day, how much protein is in their usual choices, and easy-to-consume protein-rich snacks.
Period: Overall Study
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCAs
Started | 9 | 15 | 9 | 11
Completed | 6 | 8 | 7 | 9
Not Completed | 3 | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Population: https://journals.plos.org/plosone/article/metrics?id=10.1371/journal.pone.0257742#citedHeader
Arm/Group | Intervention
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants] — Population: We had 44 participants total across four sites.
  Participants
    Arbour Trails (n = 9): number analyzed (Participants) | 9
    Arbour Trails (n = 9): <=18 years | 0
    Arbour Trails (n = 9): Between 18 and 65 years | 1
    Arbour Trails (n = 9): >=65 years | 8
    Kinnect to Wellness (n = 15): number analyzed (Participants) | 15
    Kinnect to Wellness (n = 15): <=18 years | 0
    Kinnect to Wellness (n = 15): Between 18 and 65 years | 0
    Kinnect to Wellness (n = 15): >=65 years | 15
    Village of Winston Park (n = 9): number analyzed (Participants) | 9
    Village of Winston Park (n = 9): <=18 years | 0
    Village of Winston Park (n = 9): Between 18 and 65 years | 0
    Village of Winston Park (n = 9): >=65 years | 9
    YMCA (n = 11): number analyzed (Participants) | 11
    YMCA (n = 11): <=18 years | 0
    YMCA (n = 11): Between 18 and 65 years | 1
    YMCA (n = 11): >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] — Population: Measure Analysis Population Description: We had different numbers of participants at each site, and 44 participants total across four sites.
  years
    Arbour Trails: number analyzed (Participants) | 9
    Arbour Trails | 78 [60 to 89]
    Kinnect to Wellness: number analyzed (Participants) | 15
    Kinnect to Wellness | 81 [74 to 91]
    Village of Winston Park: number analyzed (Participants) | 9
    Village of Winston Park | 84 [69 to 90]
    YMCA: number analyzed (Participants) | 11
    YMCA | 72 [62 to 91]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We had 44 participants total across four sites.
  Participants
    Arbour Trails: number analyzed (Participants) | 9
    Arbour Trails: Female | 7
    Arbour Trails: Male | 2
    Kinnect to Wellness: number analyzed (Participants) | 15
    Kinnect to Wellness: Female | 10
    Kinnect to Wellness: Male | 5
    Village of Winston Park: number analyzed (Participants) | 9
    Village of Winston Park: Female | 7
    Village of Winston Park: Male | 2
    YMCA: number analyzed (Participants) | 11
    YMCA: Female | 10
    YMCA: Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: We had 44 participants total across four sites.
  Participants
    Arbour Trail: number analyzed (Participants) | 9
    Arbour Trail: Hispanic or Latino | 0
    Arbour Trail: Not Hispanic or Latino | 9
    Arbour Trail: Unknown or Not Reported | 0
    Kinnect to Wellness: number analyzed (Participants) | 15
    Kinnect to Wellness: Hispanic or Latino | 0
    Kinnect to Wellness: Not Hispanic or Latino | 15
    Kinnect to Wellness: Unknown or Not Reported | 0
    Village of Winston Park: number analyzed (Participants) | 9
    Village of Winston Park: Hispanic or Latino | 0
    Village of Winston Park: Not Hispanic or Latino | 9
    Village of Winston Park: Unknown or Not Reported | 0
    YMCA: number analyzed (Participants) | 11
    YMCA: Hispanic or Latino | 0
    YMCA: Not Hispanic or Latino | 11
    YMCA: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Recruitment
Description: Definition: Number recruited at end of rollout. The criterion for success is to recruit 10 participants at each of 4 sites.
Time Frame: 2 month (September to October 2019)
Population: Five individuals withdrew a few days after randomization, and, since the program had not started, we recruited an additional four participants.
Measure: Number; unit: # of participants @ start of study
Groups:
- Arbour Trails: Retirement/assisted living home and independent living, Guelph, site 1
  Strength and Balance Training & Nutrition Education: Exercise:A kinesiologist-led twice-weekly program. Prior to attending the program, each attendee gets a 1:1 session with the kinesiologist to decide exercise starting levels. Group exercises start with a warm-up stepping game. Participants then perform 2 sets of 8 repetitions of each exercise, gradually progressing to an intensity of 3-8 repetitions maximum. Exercises include one each of a push, pull, squat, reach/press, lunge/step-up, lift and carry movement. After, there is a 10-minute group discussion to prompt making exercise routine at home. Nutrition:Two dietitian-led interactive group seminars to promote strategies to increase protein intake and sampling of protein-rich snacks and protein supplements. Seminar topics consider the cost to prepare high protein foods, the ability of retirement home residents to alter diet, how and why to spread protein intake through the day, how much protein is in their usual choices, and easy-to-consume protein-rich snacks.
- City of Lakes Family Health Team: Sudbury, site 2 Strength and Balance Training & Nutrition Education: Exercise:A kinesiologist-led twice-weekly program. Prior to attending the program, each attendee gets a 1:1 session with the kinesiologist to decide exercise starting levels. Group exercises start with a warm-up stepping game. Participants then perform 2 sets of 8 repetitions of each exercise, gradually progressing to an intensity of 3-8 repetitions maximum. Exercises include one each of a push, pull, squat, reach/press, lunge/step-up, lift and carry movement. After, there is a 10-minute group discussion to prompt making exercise routine at home. Nutrition:Two dietitian-led interactive group seminars to promote strategies to increase protein intake and sampling of protein-rich snacks and protein supplements. Seminar topics consider the cost to prepare high protein foods, the ability of retirement home residents to alter diet, how and why to spread protein intake through the day, how much protein is in their usual choices, and easy-to-consume protein-rich snacks.
- Village of Winston Park: Retirement/assisted living home and independent living, Kitchener, site 3
  Strength and Balance Training & Nutrition Education: Exercise:A kinesiologist-led twice-weekly program. Prior to attending the program, each attendee gets a 1:1 session with the kinesiologist to decide exercise starting levels. Group exercises start with a warm-up stepping game. Participants then perform 2 sets of 8 repetitions of each exercise, gradually progressing to an intensity of 3-8 repetitions maximum. Exercises include one each of a push, pull, squat, reach/press, lunge/step-up, lift and carry movement. After, there is a 10-minute group discussion to prompt making exercise routine at home. Nutrition:Two dietitian-led interactive group seminars to promote strategies to increase protein intake and sampling of protein-rich snacks and protein supplements. Seminar topics consider the cost to prepare high protein foods, the ability of retirement home residents to alter diet, how and why to spread protein intake through the day, how much protein is in their usual choices, and easy-to-consume protein-rich snacks.
- YMCA's: YMCA's of Cambridge and Kitchener-Waterloo, site 4
  Strength and Balance Training & Nutrition Education: Exercise:A kinesiologist-led twice-weekly program. Prior to attending the program, each attendee gets a 1:1 session with the kinesiologist to decide exercise starting levels. Group exercises start with a warm-up stepping game. Participants then perform 2 sets of 8 repetitions of each exercise, gradually progressing to an intensity of 3-8 repetitions maximum. Exercises include one each of a push, pull, squat, reach/press, lunge/step-up, lift and carry movement. After, there is a 10-minute group discussion to prompt making exercise routine at home. Nutrition:Two dietitian-led interactive group seminars to promote strategies to increase protein intake and sampling of protein-rich snacks and protein supplements. Seminar topics consider the cost to prepare high protein foods, the ability of retirement home residents to alter diet, how and why to spread protein intake through the day, how much protein is in their usual choices, and easy-to-consume protein-rich snacks.
Arm/Group | Arbour Trails | City of Lakes Family Health Team | Village of Winston Park | YMCA's
Number analyzed (Participants) | 9 | 15 | 9 | 11
# of participants @ start of study | 9 | 15 | 9 | 11

2. Primary Outcome: Feasibility - Retention
Description: Definition: Number retrained at post-rollout end. The criterion for success is 90% at rollout end.
Time Frame: Start of the program to 9 weeks
Measure: Number; unit: # of participants that completed study
Arm/Group | Arbour Trails | City of Lakes Family Health Team | Village of Winston Park | YMCA's
Number analyzed (Participants) | 9 | 15 | 9 | 11
# of participants that completed study | 6 | 8 | 8 | 9

3. Primary Outcome: Feasibility - Adherence
Description: Definition: Percentage of individuals that attended exercise and nutrition sessions.
  The criterion for success is 70% or higher.
Time Frame: 16 sessions
Measure: Mean (Full Range); unit: % of exercise sessions completed
Groups:
- Arbour Trails: Site 1
- Kinnect to Wellness: Site 2
- Winston Park: Site 3
- YMCA: Site 4
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 8 | 12 | 8 | 11
% of exercise sessions completed | 73 [62.7 to 81.6] | 66 [45.5 to 77.5] | 73 [61.5 to 82.5] | 77 [72 to 84.5]

4. Secondary Outcome: Body Weight
Description: We will measure body weight with a calibrated scale.
Time Frame: Baseline
Population: We used a standard scale to weight each participant in Kg
Measure: Mean (Standard Deviation); unit: Baseline body weight in Kg
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 9 | 15 | 8 | 11
Baseline body weight in Kg | 63.96 (12.27) | 77.09 (10.39) | 64.76 (7.63) | 66.66 (12.80)

5. Secondary Outcome: 10 Meter Walk Test
Description: Fried Frailty Index Components: walking speed via the 10-meter walk test protocol.
Time Frame: Mean change from follow up (study visit 4) and baseline
Population: 10-meter walk test protocol. (m/s)
Measure: Mean (Standard Deviation); unit: Change in gait speed (meters/second)
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 9 | 15 | 9 | 11
Change in gait speed (meters/second) | 0.08 (0.17) | 0.16 (0.24) | 0.31 (0.36) | 0.16 (0.23)

6. Secondary Outcome: Grip Strength
Description: Fried Frailty Index Components: weakness via the Jamar hand-held dynamometer
Time Frame: Mean change from follow up (study visit 4) and baseline
Population: Grip strength in Kg
Measure: Mean (Standard Deviation); unit: Change in Grip Strength (Kg)
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 9 | 12 | 9 | 11
Change in Grip Strength (Kg) | 0.17 (4.31) | -1.57 (6.24) | 0.89 (0.33) | 0.86 (6.26)

7. Secondary Outcome: 30 Second Chair Stand Test
Description: We will use a chair with a straight back without arm rests (seat 17" high), and a stopwatch. This will assess leg strength and endurance.
Time Frame: Mean change from follow up (study visit 4) and baseline
Population: Number of chair stands within 30 seconds
Measure: Mean (Standard Deviation); unit: Change number of sit to stands
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 9 | 12 | 9 | 11
Change number of sit to stands | 1.33 (2.69) | 2.44 (2.53) | 2.04 (2.45) | 0.64 (9.29)

8. Secondary Outcome: 4 Square Step Test
Description: The Four Square Step Test is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward. For older adults > 15 seconds indicates increased risk of falls
Time Frame: Mean change from follow up (study visit 4) and baseline
Population: The Four Square Step Test is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward. For older adults > 15 seconds indicates increased risk of falls
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 9 | 12 | 9 | 11
seconds | -5.14 (6.48) | 6.54 (6.15) | 5.39 (6.54) | -1.86 (3.03)

9. Secondary Outcome: EuroQol 5 Dimension Version 5-level (EQ-5D-5L)
Description: The EuroQol 5 dimension version 5-level (EQ-5D-5L) measures quality of life using 5 dimensions, on a 5 point scale, where a higher point is considered better. The scores on the subscales are given weights and summed to convert the scores to one index score. The range of possible scores for the EQ-5D-5L index is from -0.573 to 1. A higher score is better.
Time Frame: Mean change from follow up (study visit 4) and baseline
Population: Higher score is better
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCA
Number analyzed (Participants) | 9 | 15 | 9 | 11
change in score on a scale | 0.04 (0.08) | 0.06 (0.08) | 0.25 (0.33) | 0.06 (0.07)

10. Secondary Outcome: Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Description: We will use the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool to conduct interviewer administered diet recalls for 2 weekdays and 1 weekend day. Nutrient analysis is automated and will be used to quantify and compare protein and energy intakes at baseline and follow-up only. There is no scale to this section
Time Frame: Mean change from follow up (study visit 4) and baseline
Population: For protein intake at baseline, we only collected baseline measures for 40 individuals. Specific site data is not available
Measure: Mean (95% Confidence Interval); unit: protein in grams/day
Groups:
- Baseline: All sites prior to the intervention
- Follow-up: All sites after the intervention
Arm/Group | Baseline | Follow-up
Number analyzed (Participants) | 40 | 40
protein in grams/day | 69.46 [69.46 to 22.29] | 70.88 [54.80 to 77.00]
Statistical Analysis 1: Comparison: Baseline vs Follow-up; To model the interaction between exposure to the MoveStrong program and site on secondary outcomes we applied a generalized estimating equation (GEE); Test type: Other — GEE; p = 0.05, GEE; To model the interaction between exposure to the MoveStrong program and site on secondary outcomes we applied a generalized estimating equation (GEE); GEE = 1.65, 95% CI 2-sided [-4.44 to 7.73]

11. Secondary Outcome: Number of Participants With Adverse Events
Description: We will ask participants to report adverse events and falls, using Health Canada definitions. We will report serious and non-serious adverse events (total and attributable to intervention). There is no scale to this section
Time Frame: Study visit 1, 2, 3 and 4
Measure: Number; unit: participants
Groups:
- YMCAs: Site 4
Arm/Group | Arbour Trails | Kinnect to Wellness | Winston Park | YMCAs
Number analyzed (Participants) | 9 | 15 | 9 | 11
participants | 1 | 1 | 2 | 0

12. Secondary Outcome: Participant and Provider Experience
Description: We used a semi-structured interview guide to conduct exit interviews with each participant and kinesiologist. Interviews and training sessions will be audio-recorded and transcribed verbatim. Two researchers will perform thematic analyses to describe participant and provider experience and satisfaction, adaptations, and learning needs. There is no scale to this section.
Time Frame: study visit 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Over 6 months
Description: Adverse events are unfavourable or unintended occurrence in the health or well-being of a research participant; these events may or may not be related to the intervention. We reported two types of adverse events: 1) serious adverse events defined by Health Canada as "events that result in death, hospitalization, or disability", or 2) minor adverse events. We classified each adverse event as either "not related", "related", or "possibly related" to the intervention.
Groups:
- Intervention: There were two minor adverse events possibly related to the intervention and one serious adverse event related to the intervention. One participant reported groin strain while exercising but was subsequently diagnosed with hip osteoarthritis. After one-week of rest, this individual returned with a modified exercise program. The second participant had a history of right Achilles tendinitis and complained of ankle pain during the "heel drop" (i.e., impact) movement. Although all lower body exercises were ceased, after one week they withdrew from the study. One participant sustained an inferior pubic ramus fracture after a fall during the "stepping-up" movement; although this participant did not withdraw from the study, we terminated all exercises with this individual.
- Control: There were three minor and two serious adverse events not related to the intervention. One participant slipped in the living room and fractured the metatarsal bones of their left foot. Another participant fell while attempting to sit on an unlocked walker and sustained a right inferior and superior pubic ramus fracture; this participant withdrew from the study. Two participants reported to the emergency room: one with high blood pressure and the other after experiencing a transient ischemic attack. The last participant was at home when they experienced a seizure due to unknown causes and was admitted to the hospital for observation. The participants that experienced the pubic ramus fractures and the seizure were categorized as serious adverse events as a result of being hospitalized.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/44 | 2/44
Other Adverse Events (participants affected / at risk) | 0/44 | 3/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=44) | Control (N=44)
Intervention (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — One participant slipped in the living room and fractured the metatarsal bones. Another fell while sitting on an unlocked walker and sustained a right inferior and superior pubic ramus fracture. One sustained an inferior pubic ramus fracture.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=44) | Control (N=44)
Cardio (Cardiac disorders) | 0 (0) | 3 (3) — high blood pressure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT04037436/Prot_SAP_ICF_000.pdf